CLINICAL TRIAL: NCT05252000
Title: Clinical and Microbiologic Outcomes of Adjunctive Antimicrobial Photodynamic Therapy in the Non-surgical and Surgical Treatment of Teeth With Periodontal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shreena Pranav Bhakta, resident, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-DB-21-0998
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Periodontal Diseases
Keywords: plaque; laser therapy
MeSH Terms: conditions — Periodontal Diseases; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- mechanical debridement and adjunctive aPDT (Experimental)
  Interventions: Device: mechanical debridement; Device: adjunctive aPDT
- mechanical debridement and sham aPDT (Active Comparator)
  Interventions: Device: mechanical debridement; Device: sham aPDT

INTERVENTIONS:
Device: mechanical debridement — subjects will receive traditional non-surgical mechanical debridement of tooth surfaces with scalers and ultrasonics removing supragingival and subgingival plaque
Device: adjunctive aPDT — Antimicrobial photodynamic therapy will be done at tooth sites by applying a photosensitizing dye methylene blue (0.1mg/ml) with a disposable syringe from the bottom of pocket in a coronal direction. After 3 minutes in situ, the surrounding gingival tissues will be irradiated at six sites around the tooth using a diode laser with a wavelength of 660nm, providing an energy density of 10 J/site, 100mW power, time equal to 100 seconds. After irradiation, the site will be thoroughly rinsed with saline.
  Arms: mechanical debridement and adjunctive aPDT
Device: sham aPDT — subjects will receive saline and non-light emitting laser on the tooth
  Arms: mechanical debridement and sham aPDT

SUMMARY:
The purpose of this study is to compare clinical outcomes after mechanical debridement of at sites exhibiting plaque induced inflammation with or without adjunctive Antimicrobial photodynamic therapy (aPDT) and to assess the the microbiologic profile before and after treatment with or without aPDT

ELIGIBILITY:
Inclusion Criteria:

* One pocket on each side of the mouth (split design)
* Single rooted tooth
* Pocket depths measured greater than 4mm with bleeding on probing
* Horizontal bone loss
* No furcation involvement

Exclusion Criteria:

* current heavy smokers (>10 cigarettes/day)
* have uncontrolled diabetes (HbA1c ≥ 6.5%)
* other uncontrolled systemic diseases that may comprise healing, such as Vitamin C deficiency, any neutrophil deficiencies, immunodeficiency syndromes, or leukemia
* taking antibiotics within 3 months before the procedure
* vertical bone defects that requires surgical regenerative treatment.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of bleeding sites (Bleeding On Probing) | baseline, at the re-evaluation appointment(4 to 6 weeks after baseline), and 3 months after the osseous surgery
  Bleeding on probing will be evaluated by gently sweeping the periodontal probe just within the gingival sulcus of the tooth and the presence or absence of bleeding will be recorded.
Change in probing depth (Periodontal pocket depth ) | baseline, at the re-evaluation appointment (4 to 6 weeks after baseline), and 3 months after the osseous surgery
  Periodontal pocket depth is measured from the free gingival margin to the base of the pocket, with a UNC periodontal probe with 1mm measurement units

SECONDARY OUTCOMES:
change in microbiologic profile of plaque | baseline, at the re-evaluation appointment(4 to 6 weeks after baseline), and 3 months after the osseous surgery
  Plaque sampling will be performed using a curette within the gingival sulcus of the inflamed site. The sample sites will first be isolated by cotton rolls and supragingival and marginal plaque will be removed before subgingival biofilm samples collected using sterile scalers. The collected samples will be immediately placed in separate sterile Eppendorf tubes containing 0.15 ml TE .Samples will be stored at -80 °C until further analysis.
change in microbiologic profile of gingival crevicular fluid(GCF) | baseline, at the re-evaluation appointment(4 to 6 weeks after baseline), and 3 months after the osseous surgery
  GCF will be collected from the sulcus around the target tooth using paper strips (PerioPaper, Oraflow). With proper isolation using cotton rolls in the buccal and lingual aspects of the study site, the area will be dried for 5 seconds with compressed air. The paper strip will be gently introduced into the mucosal crevice around the tooth for 30 seconds per site in four sites.The strips will then be removed from the crevice, and the volume of fluid collected in each strip measured using a micromoisture metering device (Peritron, Oraflow). After confirming the adequateness of the volume, the paper strips from each tooth will be transferred into labeled tubes and stored at -80 C for later use. For analysis, the paper strips will be analyzed using multiplexed fluorescent bead-based immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Shreena P Bhakta, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No